CLINICAL TRIAL: NCT06280274
Title: Perioperative Metformin Use in Patients Undergoing Total Joint Replacement Surgery: A Pilot Study
Brief Title: Metformin Use in Patients Undergoing Total Joint Replacement Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Ryland Kagan, Assistant Professor of Orthopaedics and Rehabilitation, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00025798
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-08

CONDITIONS: Hyperglycemia
Keywords: Arthroplasty; Hip; Knee; Metformin; glycemic variability
MeSH Terms: conditions — Hyperglycemia | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Oral metformin hydrochloride
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin 500mg oral once daily for 7 days, increased to 1000mg (500mg twice daily) for another 7 days, taken in morning and evening with meals, for a total of 14 days of treatment prior to surgery. Continue dose on day of surgery and up to post operative day 2, or until time of discharge, whichever happens first.
  Arms: Treatment
Other: Placebo — Placebo tablet
  Arms: Placebo

SUMMARY:
The goal of this pilot, randomized, single-blind, placebo-controlled trial is to evaluate the feasibility of and provide preliminary information for a multi-center randomized controlled trial that will assess the effects of metformin on blood sugar control in patients after total hip or total knee replacement surgery.

The primary objective of this study is to assess the feasibility of conducting a large, randomized trial with regards to timely recruitment, study drug administration, protocol adherence, and overall retention in patients undergoing total joint arthroplasty.

Secondarily, the investigators aim to obtain preliminary estimates of group-specific outcome means and variances for primary and secondary outcomes of a larger future trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18-99 years
* Undergoing total hip or total knee arthroplasty, including elective, primary, and revision surgeries
* Ability to take oral medication and be willing to adhere to the prescribed metformin regimen regardless of current, past, or no metformin use.

Note: Patients with or without type 2 diabetes are considered eligible. (E.g.)

* Type 2 diabetic on metformin
* Type 2 diabetic on metformin and other medication, including insulin
* Type 2 diabetic on medication but not metformin
* Pre-diabetic
* Non-diabetic

Exclusion Criteria:

* Advanced renal insufficiency (glomerular filtration rate (GFR) < 45, or chronic kidney disease (CKD) stage 3B or higher)
* Advanced liver cirrhosis or failure (Child-Pugh class B or C)
* Congestive heart failure (New York Heart Association (NYHA) class 3 or 4)
* Current alcohol abuse within 30 days of surgery (>4 standard servings daily for men, >3 standard servings daily for women)
* Type 1 diabetes
* Received contrast dye within 48 hours of surgery
* Vulnerable populations: Children, pregnant women, neonates, decisionally impaired adults, prisoners

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Rate of participant enrollment | 3 months
  Feasibility defined by an average of four participants per month successfully enrolled and randomized.
Rate of appropriate study drug administration | 3 months
  Feasibility defined by ≥90% participants receiving 1000mg metformin or placebo daily by day of surgery, assessed via combination of self-report and counting of remaining tablets.
Rate of participant adherence to trial intervention per protocol | 3 months
  Feasibility defined by ≥90% participant adherence to trial intervention per protocol.
Rate of participant retention to 90-day follow up | 3 months
  Feasibility defined by ≥90% retention to follow up at 90 days.

SECONDARY OUTCOMES:
Perioperative glycemic variability | 3 months
  Defined as coefficient of variation (CV) = standard deviation / mean of blood glucose levels
Sliding scale insulin utilization | 3 months
  Measured by total number of units administered from time of surgery to discharge.
Hospital length of stay | 3 months
  Measured in days.
90-day Rate of surgical site infection | 3 months
  Defined by criteria published by Centers for Disease Control and Prevention.
90-day Rate of periprosthetic joint infection | 3 months
  Defined by criteria published in 2018 by Musculoskeletal Infection Society (MSIS).
90-day Rate of mortality | 3 months
90-day rate of readmission | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ryland Kagan, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morrell A, Shelofsky S, Hoffman H, McCallister C, Huff TW, Schabel KL, O'Glasser AY, Kagan RP. Perioperative metformin use in patients undergoing total joint replacement surgery: protocol for a randomised, placebo-controlled pilot study. BMJ Open. 2025 Apr 8;15(4):e091446. doi: 10.1136/bmjopen-2024-091446. PMID 40204318
- See also: Metformin labeling — https://www.accessdata.fda.gov/drugsatfda_docs/label/2017/020357s037s039,021202s021s023lbl.pdf